CLINICAL TRIAL: NCT00926458
Title: NON-Invasive Examinations of Coronary Artery Disease
Acronym: NONCAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herning Hospital (Other)
Responsible Party: Ole May, Cardiovascular Research Unit, Region Hospital Herning
Other Study IDs: NONCAD
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Artery Disease
Keywords: stress echocardiography; coronary angiography; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to evaluate and compare the value of 5 different non-invasive diagnostic methods in patients with chest pain suspected for coronary artery disease. The investigators intend to include 200 patients over a 3 year period in the study. The participants will be recruited from patients referred to coronary angiography at the institution. Before the angiography the participants will (1) test the effect of sublingual Nitroglycerin, (2) give their medical history so mathematical models can estimate the probability of the presence of coronary artery disease, (3) take part in a contrast stress echocardiography and (4) a 2D-strain stress echocardiography and a myocardial scintigraphy. Stenosis found at the angiography will be the gold standard.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the diagnostic value of various non-invasive methods. The study is divided into five substudies:

Substudy NITRO

Purpose: To investigate whether a subjective effect of Nitroglycerine is associated with significantly narrowed coronary arteries.

The participants are instructed to alternate between rest and Nitroglycerine as treatment for chest pain attacks during a 2 week period. Chest pain score is recorded in a diary handed out at day 1 together with 30 tablets Nitroglycerine in the maximal tolerated dose.

Substudy SCORE

Aim: To test and compare the ability of different statistical methods using clinical data to predict the presence of narrowed coronary arteries in a contemporary Danish population.

Substudy CONTRAST

Aim: To evaluate if the blood flow in an area in the heart muscle measured by contrast adenosine stress echocardiography can predict the presence of significant stenosis in the coronary artery supplying the area.

Substudy 2D strain

Aim: To Evaluate if lack of increase in 2D strain during adenosine stress echocardiography can predict the presence of narrowed coronary arteries.

Substudy SPECT

Aim: To evaluate whether the result of a myocardial scintigraphy can predict symptomatic chest pain relief 6 months after a coronary angiography and possible treatment with balloon or bypass surgery.

Participants: Annually around 1,500 coronary angiographies are performed at Region Hospital Herning. We intend to include 200 patients referred by their physicians to coronary angiography in the study and expect the data collection phase to last 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Intermittent episodes of chest pain (more than two attacks, minimum one attack/week)
2. Signed written informed consent
3. Sinus rhythm (ECG)
4. Age above 18 years

Exclusion Criteria:

1. Previously (known) myocardial infarction or unstable angina with dynamic changes in the ECG or biomarkers (serology)
2. CA performed earlier in life
3. Known significant cardiac valve disease
4. Asthma (not COPD)
5. Incapable of performing an exercise test
6. Malignant Disease
7. Senile dementia or other conditions causing impaired cooperation
8. Previous participation in the project
9. NTG intolerance
10. Pregnancy
11. Bundle branch block (QRS > 120 ms)
12. ECG changes:

    * Pathologic Q-wave in at least two leads:
    * QS-complex or Q-wave > 0.02 sec. in V2-V3
    * QS-complex or Q-wave > 0.03 sec. and > 0.1 mV in I, II, aVL, aVF or V4-V6
    * Pathologic negative T-wave (in V3-6 and I, II) unless this is part of a left ventricular hypertrophy and strain pattern
13. Brady pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for coronary angiography at Region Hospital Herning are screened for the study and all patients complying with the in-/exclusion criteria are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ole May, MD, Ph.D., Principal Investigator — Cardiovascular Research Unit
Locations (1):
- Cardiovascular Research Unit, Regionhospital Herning, Herning, Denmark